CLINICAL TRIAL: NCT04709666
Title: Difficult Biliary Cannulation in Patients With Distal Malignant Biliary Obstruction: an Underestimated Problem
Acronym: DBC 01
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2143-2
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Biliary Condition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endsocopic Retrograde ColangioPancreatography (ERCP): Endsocopic Retrograde ColangioPancreatography (ERCP)
  Interventions: Procedure: Endsocopic Retrograde ColangioPancreatography (ERCP)

INTERVENTIONS:
Procedure: Endsocopic Retrograde ColangioPancreatography (ERCP)

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is the primary therapeutic procedure for many bilio-pancreatic diseases, and requires the first crucial step of the successful deep cannulation of the common bile duct through the Vater's papilla. Difficult biliary cannulation (DBC) is a well-recognized risk factor for adverse events (AE) and cannulation failure, which has been reported in about 11% of ERCP regardless of their indication and a relevant heterogeneity in definition of DBC is present in the available studies. More recently, DBC during ERCP has been precisely defined by the European Society of Gastrointestinal Endoscopy (ESGE) as follows: more than 5 contacts with the papilla whilst attempting to cannulate; more than 5 minutes spent attempting to cannulate after visualization of the papilla; more than one unintended pancreatic duct cannulation or opacification (4). To date, the rate of DBC has not been calculated for specific sub-groups of ERCP indications. In particular, the rate of DBC in the setting of distal malignant biliary obstruction (DMBO), a frequent indication for ERCP, has not yet been described. DMBO is generally secondary to pancreatic adenocarcinoma, distal cholangiocarcinoma, ampullary carcinomas or adenopathy/metastasis from other cancers, and could potentially increase the complexity of the procedure as the tumor compression or infiltration alter the normal duodenal/papillary anatomy or determine duodenal rigidity.

In this study, we aimed to investigate the rate of DBC and the outcome of patients undergoing ERCP for DMBO.

ELIGIBILITY:
Inclusion Criteria:

* With an age above or equal to 18,
* From which informed consent has been obtained,
* patients undergoing ERCP carried out by expert operators for DMBO due to pancreatico-biliary malignancies.

Exclusion Criteria:

- Patients who do not meet all of the listed inclusion criteria will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be recruited at the UO of Gastroenterology and digestive endoscopy of the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of DBC | 6 Months
  To investigate the rate of DBC and the outcome of patients undergoing ERCP for DMBO.

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No